CLINICAL TRIAL: NCT06079424
Title: Risk Markers of Arterial Aging and Subsequent Risk of Cardiovascular Diseases and Beyond. The Paris Prospective Study III-2
Brief Title: Risk Markers of Arterial Aging. The Paris Prospective Study III-2
Acronym: PPS3-2
Status: Recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C21-67
Record Dates: First submitted 2023-09-26; First posted 2023-10-12 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Arterial Stiffness
Keywords: risk factors; cohort; cardiovascular diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — EDTA and citrate plasmatic samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Level of vascular aging: community-based prospective longitudinal cohort
  Interventions: Other: high-precision carotid echo-tracking

INTERVENTIONS:
Other: high-precision carotid echo-tracking — evaluation of vascular aging parameters and baroreflex sensitivity

SUMMARY:
The main objectives of PPS3-2 are (i) to describe the dynamics of vascular aging and baroreflex sensitivity 12 to 16 years a part, (ii) to identify their determinants, and (iii) to quantify the subsequent risk of cardiovascular diseases.

DETAILED DESCRIPTION:
Since May 2008, PPS3 is being following the CVD morbidity of 10157 healthy volunteers aged 50-75 years at baseline. In PPS3-2, we plan to re-invite survivors and volunteers of PPS3 to undergo a second physical examination. In particular, they will undergo a second high-precision carotid echotracking to measure vascular aging parameters and baroreflex sensitivity, permitting to study their respective dynamics. They will also underwent for the first time ultra fast echo of the radial artery to measure vascular aging parameters of the medium-sized arteries. According to fundings, blood samples will be taken and stored at -80°C in the whole population or in a subsample.

ELIGIBILITY:
Inclusion Criteria:

* Being enrolled in PPS3 and having signed an informed consent for PPS3-2

Exclusion Criteria:

* Institutionalized participants
* Participants under guardianship
* Participants under judicial safeguard measure

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and women aged 60 to 95 years who are participants of the PPS3 study and have accepted to undergo a second physical examination and answer to health questionnaires in primary care health centre in Paris that is subsidized by the French Health Insurance System.
Sampling Method: Non-Probability Sample
Enrollment: 7500 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2031-05 (Estimated); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
carotid diameter | by 2027
  high precision carotid echo tracking diameter in mm
intima media thickness | by 2027
  high precision echo tracking intima media thickness of the common carotid artery in mm
carotid plaques | by 2027
  high precision carotid echo tracking carotid plaques
wall cross sectional area | by 2027
  high precision carotid echo tracking carotid wall cross sectional area, mm2
distensibility coefficient | by 2027
  high precision carotid echo tracking distensibility coefficient in 10-3/kPa
elastic modulus | by 2027
  high precision carotid echo tracking Young's elastic modulus, 10-3*kPa
pulse wave velocity | by 2027
  high precision carotid echotracking pulse wave velocity, m/s
carotid wall stress | by 2027
  high precision carotid echotracking circumferential wall stress in kPa
stiffness | by 2027
  high precision carotid echotracking Beta stiffness index
pulse pressure | by 2027
  high precision carotid echotracking pulse pressure in mmHg

SECONDARY OUTCOMES:
brachial artery diameter | by 2027
  ultra high frequency ultrasound radial artery diameter in mm
thickness of the intima media of the radial artery | by 2027
  ultra high frequency ultrasound radial artery intima media thickness in mm
arterial plaques | by 2027
  ultra high frequency ultrasound radial artery plaques
wall cross sectional area of the radial artery | by 2027
  ultra high frequency ultrasound radial artery wall cross sectional area, mm2
distensibility of the radial artery | by 2027
  ultra high frequency ultrasound radial artery distensibility coefficient in 10-3/kPa
elastic modulus of the radial artery | by 2027
  ultra high frequency ultrasound radial artery Young's elastic modulus, 10-3*kPa
pulse wave velocity of the radial artery | by 2027
  ultra high frequency ultrasound radial artery Pulse wave velocity, m/s
stiffness index of the radial artery | by 2027
  ultra high frequency ultrasound radial artery Beta stiffness index
wall stress of the radial artery | by 2027
  ultra high frequency ultrasound radial artery Circumferential wall stress, kPa
pulse pressure of the radial artery | by 2027
  ultra high frequency ultrasound radial artery Pulse Pressure, mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe Empana, MD, PhD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Centre d'Investigation Précliniques, Paris, France

IPD SHARING:
Plan to Share IPD: No